CLINICAL TRIAL: NCT01379170
Title: Effects of Thyroid Hormone Treatment on Mitochondrial Function, Ectopic Fat Accumulation, Insulin Sensitivity and Brown Adipose Tissue in Type 2 Diabetes Mellitus
Brief Title: Thyroid Study Type 2 Diabetes Mellitus (T2DM)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MEC10-3-085
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes; Hypothyroidism
Keywords: brown adipose tissue; mitochondrial dysfunction; insulin resistance
MeSH Terms: conditions — Diabetes Mellitus; Hypothyroidism; Mitochondrial Diseases; Insulin Resistance | interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Type 2 diabetes, de novo hypothyrodism treatment (Experimental): Type 2 diabetic patients with de novo hypothyroidism will be included in this arm and will receive 3 months of treatment with Euthyrox (standard protocol).
  Interventions: Drug: Euthyrox (levothyroxine)

INTERVENTIONS:
Drug: Euthyrox (levothyroxine) — A dose of 25 μg per day of Euthyrox® will be administered orally during the first week and will be increased to 50 μg per day during the second week and to 75-100 μg per day in the third week depending on TSH, free T4 and T3 concentrations monitored throughout the treatment period. Patients will be instructed to take Euthyrox® after an overnight fast, 30 min before breakfast in the morning daily. After 3 months, free T4 and total T3 concentration must be in the normal range (free T4: 8.0-26 pmol/l, T4: 60-140 nmol/l and T3 1.2 - 3.4 nmol/l) and TSH 0.4-2.5 mU/l.
  Other Names: Euthyrox/levothyroxine

SUMMARY:
Background of the study:

Thyroid hormones, thyroxine (T4) and triiodothyronine (T3), are known to promote weight loss, which could be beneficial for treating obesity, and type 2 diabetes. Thyroid hormone treatment stimulates energy expenditure resulting in increased body heat production, in which brown adipose tissue play an important role. It is hypothesized that thyroid hormones would induce increased energy expenditure via a process called mitochondrial uncoupling, thereby creating an inefficient energy status. Indeed, an in vivo study showed a 70% increased flux through the tricarboxylic acid cycle (TCA) and an unchanged ATP synthesis rate upon T3 treatment in lean, healthy young men. The disproportionate increase in TCA flux compared with ATP synthesis suggests increased mitochondrial uncoupling. It is however unknown whether increased mitochondrial uncoupling would increase fat oxidation and exerts favorable effects on insulin sensitivity. There is compelling evidence that type 2 diabetic patients have high levels of fat accumulation in non-adipose tissues, such as skeletal muscle, heart and liver. Ectopic fat accumulation is related to insulin resistance, however, why this fat accumulates in peripheral organs is not known. Recently, studies reported compromised mitochondrial oxidative capacity in type 2 diabetic patients and first-degree relatives of diabetic patients, suggested to play an important role. Therefore, subjects suffering from overweight and/or type 2 diabetes with overt hypothyroidism form an interesting group for examining the metabolic effects of thyroid hormone treatment, as less is known about the effects of thyroid hormone treatment in these groups.

Objective of the study:

The purpose of this study is to evaluate whether thyroid hormone replacement therapy in type 2 diabetic patients suffering from overt hypothyroidism, will improve muscular mitochondrial function, lower ectopic fat accumulation in muscle and liver, increase brown adipose tissue activity and enhance insulin sensitivity.

Study design:

Type 2 diabetic patients diagnosed with hypothyroidism will undergo 3 months of thyroid hormone replacement therapy (THRT) (Euthyrox®, Merck, Germany). Patients will be metabolically characterized (such as insulin sensitivity and fat accumulation in peripheral tissues) before and after this thyroid hormone replacement therapy.

Study population:

17 type 2 diabetic patients diagnosed with overt hypothyroidism (9 from the Netherlands, 8 from Germany which will only do the PET-CT)

Primary study parameters/outcome of the study:

Thyroid hormone-induced change in whole body insulin sensitivity (change in insulin-stimulated glucose disposal) and muscle mitochondrial function.

Secondary study parameters/outcome of the study (if applicable):

Thyroid hormone-induced change of lipid content in skeletal muscle and liver and brown adipose tissue activity.

ELIGIBILITY:
Inclusion Criteria:

* Male or postmenopausal females
* Age 40-65 years
* Body mass index (BMI) < 40 and > 27 kg/m2
* Stable dietary habits (no weight loss/gain >3 kg in the last 6 months)
* Stable physical activity levels for at least six months
* Newly diagnosed hypothyroid, non-insulin dependent type 2 diabetic patients having TSH values higher then > 4.0 mU/l and lowered concentrations of free T4 < 8.0 pmol/l.
* Type 2 diabetic patients using sulphonylurea and or metformin therapy for at least six months with a constant dose for at least two months.
* Hypothyroid diabetic patients due to Hashimoto disease (TPO > 100 IE/ml; Tg > 344 IE/ml), should have no auto-antibodies against glutamic acid decarboxylase (GAD), IA-2 and insulin to exclude type 2 polyglandular autoimmune syndrome (PGAII) (to exclude type 1 diabetes).
* Type 2 diabetic patients should have a HbA1c level < 8.0%
* Type 2 diabetic patients will be included when having no diabetes-related co-morbidities like cardiovascular diseases, diabetic foot, polyneuropathy, retinopathy.

Exclusion Criteria:

* Unstable body weight
* Participation in an intensive weight-loss program or vigorous exercise program during the last year before the start of the study
* Medical history including active cardiovascular disease, i.e. history of coronary artery disease (i.e. history of angina pectoris, percutaneous transluminal coronary angioplasty or coronary artery bypass grafting) or cardiac arrhythmias.
* Liver disease or liver dysfunction (ALT>2.5 x increased)
* Impaired renal function (creatinine > 120 umol/L)
* Systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg
* Hb <7.4 mmol/l (12 g/dl) in women, and <8.1 mmol/l (13 g/dl) in men
* Abuse of drugs and/or alcohol
* Contraindications for MRI scanning (please see appendix III: MRI contraindication questionnaire)
* Patients with history of thyroid cancer
* Patients using α and/or β blockers
* Severe diabetes which requires application of insulin or patients with diabetes-related complications
* History of psychiatric disease
* Diabetes related co-morbidities like cardiovascular diseases, diabetic foot, polyneuropathy, retinopathy.
* Use of medications known to interfere with glucose homeostasis (i.e. corticosteroids, thiazolidinediones)
* Hypothyroid diabetic patients due to Hashimoto disease with positive test values for auto-antibodies against GAD, IA-2 and insulin to exclude type 1 diabetes.
* Use of anticoagulants, other than platelet aggregation inhibitors.
* Patients that have donated blood in the past 6 months

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Thyroid hormone-induced change in whole body insulin sensitivity (change in insulin-stimulated glucose disposal) and muscle mitochondrial function | 3 months
  see title

SECONDARY OUTCOMES:
Thyroid hormone-induced change of lipid content in skeletal muscle and liver and brown adipose tissue activity | 3 months
  see title

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands